CLINICAL TRIAL: NCT07066176
Title: Development of Intestinal Permeability Tests for Clinical Nutrition and Metabolic Health Studies
Brief Title: Establishing and Validating a Meal-provoked Intestinal Permeability Test for Nutritional and Metabolic Health Clinical Research.
Acronym: Gut-Perm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Alain Veilleux, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025-178
Record Dates: First submitted 2025-06-30; First posted 2025-07-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Intestinal Permeability
Keywords: intestinal permeability
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water (No Intervention): Mannitol and lactulose diluted in water (500mL)
- Mixed meal beverage (Placebo Comparator): Mannitol and lactulose diluted in mixed meal beverage (500mL)
  Interventions: Dietary Supplement: Mixed meal beverage
- Mixed meal beverage and aspirin (Experimental): Aspirin (650mg) prior to mannitol and lactulose diluted in mixed meal beverage (500mL)
  Interventions: Drug: Aspirin; Dietary Supplement: Mixed meal beverage

INTERVENTIONS:
Drug: Aspirin — Aspirin 650mg prior mixed meal beverage
  Arms: Mixed meal beverage and aspirin
Dietary Supplement: Mixed meal beverage — Mixed meal beverage
  Arms: Mixed meal beverage; Mixed meal beverage and aspirin

SUMMARY:
Development of Intestinal Permeability Tests for Clinical Nutrition and Metabolic Health Studies

DETAILED DESCRIPTION:
Crossover clinical trial on 10 subjects (5 women, 5 men) with 3 intestinal permeability tests (3-day washout) as follows: 1) fasting; 2) meal-provoked; and 3) meal-provoked with acute aspirin challenge to assess the test's feasibility and capacity to detect alterations in intestinal permeability after aspirin-induced intestinal barrier defects.

Each test will be performed after a 12h fast. Subjects will provide fasting blood and urine samples, fully empty their bladders and drink 50mL of water with/without soluble aspirin (650mg). After 30 min., subjects will drink 500mL of water or mixed meal beverage (22g protein, 26g fat, 52g carbs) with mannitol (2g) and lactulose (4g). A standardized snack and water (200mL) will be provided at 3h. Blood samples will be taken at 2h, 3h and 4h. All urine will be collected over 5 hours. Collection times were adapted to account for potential delays in gastric emptying (mixed meal vs. water). Lactulose-to-mannitol ratios, by HPAEC-PAD method, in urine and blood will be compared by phases using mixed linear models.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18-65y
* BMI <40

Exclusion Criteria:

* Enteropathies
* Food intolerance or allergy related to the protocol
* Pregnancy or breastfeeding within the last 3 months
* Contraindications for aspirin - see Monograph

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Intestinal permeability | From baseline to hour 5
  lactulose-to-mannitol ratio in urine

SECONDARY OUTCOMES:
Intestinal permeability | At baseline, hour 2, hour 3 and hour 4
  lactulose-to-mannitol ratio in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Alain Veilleux, PhD, Principal Investigator — Laval University
Locations (1):
- INAF, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No